CLINICAL TRIAL: NCT01672320
Title: Outcomes of Robotic Total Hip Arthroplasty: A Prospective Study
Brief Title: Outcomes of Robotic Total Hip Arthroplasty
Status: Withdrawn | Type: Observational
Why Stopped: No patients will be recruited at Massachsetts General hospital. IRB approval changed to core center.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: MAKO Surgical Corp. (Industry)
Responsible Party: Principal Investigator, Charles R. Bragdon, Research Scientist, Massachusetts General Hospital
Other Study IDs: 2012P000809
Record Dates: First submitted 2012-08-10; First posted 2012-08-24 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis
Keywords: Robotic; Arthroplasty; Total Hip Arthroplasty; Cup Positioning; Outcomes
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phase II: An evaluation of long-term outcomes, patient reported outcomes, and radiographic analysis will be conducted prospectively on 500 patients
- Phase I: An analysis of post-operative component positioning will be evaluated for 500 patients, retrospectively.

SUMMARY:
The objectives of this study are to evaluate the clinical value of robotic-assisted total hip arthroplasty with respect to acetabular cup implantation, and to document the long-term clinical outcome of patients with Total Hip Arthroplasty (THA). IRB approval will be obtained at every study site to evaluate the basic clinical outcomes and post-operative component placement accuracy of each MAKO® THA patient.

The hypothesis is that robotic preparation of the acetabulum will significantly reduce the variability and inaccuracy in the component alignment parameters that lead to post-operative complications, including implant failure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 20 to 75 years of age
* Subjects requiring primary total hip replacement
* Contralateral hip should be relatively free from arthritis for comparison purposes, specifically with less than a grade of 2 on the Kellgren-Lawrence Scale.
* Subjects diagnosed with osteoarthritis or traumatic arthritis
* Subjects with avascular necrosis
* Subjects who demonstrate the ability to return for follow-up for the next 10 years

Exclusion Criteria:

* Subjects with difficulty understanding protocol for any reason
* Subjects with a limited life span
* Subjects with inflammatory hip disease, previous joint infection, or those requiring hip revision surgery
* Female subjects who are pregnant, or who plan to get pregnant while enrolled in the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults requiring a total hip arthroplasty procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Survivorship of Components | 10 Years
  Defined as implant remaining in subject.
Adverse Events | 10 Years
  Protocol deviations, complications, "lost to follow-up"

SECONDARY OUTCOMES:
Retrieval Analysis of implants from revision surgery | Up to 10 Years
  When possible, analysis of the THR components that are removed at revision surgery will be anlaysed for signs of component impingment or signs of damage related to component position. These observations will be correlated to the clinical reason for revision.

OTHER OUTCOMES:
Assessment/questionaire HOOS | Pre-op, 1, 3, 5, 7, 10 years after surgery
  Hip Disability and Osteoarthritis Outcome
Assessment/Questionaire UCLA Activty Score | Pre-op, 1, 3, 5, 7, 10 years after surgery
  Assesses level of activity
Assessment/Questionaire EQ-5D | Pre-op, 1, 3, 5, 7, 10 years after surgery
  General health and cost effective analysis
Assessment/questionaire | Pre-op, 1, 3, 5, 7, 10 years after surgery
  Hip desease specific questionaire
Assessment/Questionaire Case Mix Indicator | Pre-op, 1, 3, 5, 7, 10 years after surgery
  Identifies comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States